CLINICAL TRIAL: NCT03103204
Title: Clinical, Microbial and Biochemistry Evaluation of Obese Individuals Submitted to One-stage Full-mouth Disinfection. A Clinical Control Parallel Study
Brief Title: Treatment of Periodontitis in Obese Individuals
Acronym: CLIMBEO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Taubate (Other)
Responsible Party: Principal Investigator, Jose Roberto Cortelli, Head of Periodontics Department, University of Taubate
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTaubate
Record Dates: First submitted 2017-03-14; First posted 2017-04-06 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Obese; Obesity, Morbid; Periodontitis
Keywords: Obesity; Periodontitis; Therapeutics; Chlorhexidine
MeSH Terms: conditions — Obesity; Obesity, Morbid; Periodontitis | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Normal weight full-mouth disinfection (Experimental): * Normal weight (body mass index 18.5 - 24.9 kg/m2) individuals with chronic periodontitis
  * Full-mouth manual scaling and root planing within 24 hours
  * tongue cleaning with chlorhexidine gel 1% for 1 minute
  * tonsils disinfection with chlorhexidine spray 0.2%
  * rinsing with 15mL of 0.2% chlorhexidine solution for 30 seconds before and after dental scaling
  * subgingival irrigation of all periodontal pockets with 1% chlorhexidine solution
  * daily rinsing with 0.2% chlorhexidine solution (15mL/30 seconds/2 times a day
  Interventions: Combination Product: One-stage full-mouth disinfection with chlorhexidine
- Overweight full-mouth disinfection (Experimental): * Overweight (body mass index 25.0 - 29.9 kg/m2) individuals with chronic periodontitis
  * Full-mouth manual scaling and root planing within 24 hours
  * tongue cleaning with chlorhexidine gel 1% for 1 minute
  * tonsils disinfection with chlorhexidine spray 0.2%
  * rinsing with 15mL of 0.2% chlorhexidine solution for 30 seconds before and after dental scaling
  * subgingival irrigation of all periodontal pockets with with 1% chlorhexidine solution
  * daily rinsing with 0.2% chlorhexidine solution (15mL/30 seconds/2 times a day
  Interventions: Combination Product: One-stage full-mouth disinfection with chlorhexidine
- Obesity I full-mouth disinfection (Experimental): * Obesity I (body mass index 30.0 - 34.9 kg/m2) individuals with chronic periodontitis
  * Full-mouth manual scaling and root planing within 24 hours
  * tongue cleaning with chlorhexidine gel 1% for 1 minute
  * tonsils disinfection with chlorhexidine spray 0.2%
  * rinsing with 15mL of 0.2% chlorhexidine solution for 30 seconds before and after dental scaling
  * subgingival irrigation of all periodontal pockets with with 1% chlorhexidine solution
  * daily rinsing with 0.2% chlorhexidine solution (15mL/30 seconds/2 times a day
  Interventions: Combination Product: One-stage full-mouth disinfection with chlorhexidine
- Obesity II full-mouth disinfection (Experimental): * Obesity II (body mass index 35.0 - 39.9 kg/m2) individuals with chronic periodontitis
  * Full-mouth manual scaling and root planing within 24 hours
  * tongue cleaning with chlorhexidine gel 1% for 1 minute
  * tonsils disinfection with chlorhexidine spray 0.2%
  * rinsing with 15mL of 0.2% chlorhexidine solution for 30 seconds before and after dental scaling
  * subgingival irrigation of all periodontal pockets with with 1% chlorhexidine solution
  * daily rinsing with 0.2% chlorhexidine solution (15mL/30 seconds/2 times a day
  Interventions: Combination Product: One-stage full-mouth disinfection with chlorhexidine
- Obesity III full-mouth disinfection (Experimental): * Obesity III (body mass index ≥ 40.0 kg/m2) individuals with chronic periodontitis
  * Full-mouth manual scaling and root planing within 24 hours
  * tongue cleaning with chlorhexidine gel 1% for 1 minute
  * tonsils disinfection with chlorhexidine spray 0.2%
  * rinsing with 15mL of 0.2% chlorhexidine solution for 30 seconds before and after dental scaling
  * subgingival irrigation of all periodontal pockets with with 1% chlorhexidine solution
  * daily rinsing with 0.2% chlorhexidine solution (15mL/30 seconds/2 times a day
  Interventions: Combination Product: One-stage full-mouth disinfection with chlorhexidine

INTERVENTIONS:
Combination Product: One-stage full-mouth disinfection with chlorhexidine — Mechanical procedures, composed of full-mouth dental scaling and root planning and dental prophylaxis, will be completed within 24 hours (2 appointments in 2 consecutive mornings or afternoons).
  Chlorhexidine will be used as the antimicrobial agent in different concentrations (0.2%, 1% and 2%) and vehicles (solution, gel).
  Oral hygiene instructions will be given for all participants.

SUMMARY:
Obesity and gum diseases are highly prevalent in all parts of the world. Obesity can negatively influence severity and progression rates of gum diseases. Presence of fat in the body determines a general systemic state of inflammation. On the other hand, when gum diseases are successfully treated systemic and local inflammation decrease. In addition reductions in glycemic blood levels are also observed after treatment. Periodontitis is one type of gum disease that is associated with bone loss. It could be treated within 24 hours by using a protocol, which combines dental debridement and mouthwash. This treatment protocol, named "one-stage full-mouth disinfection" works well in individuals of normal weight. However, there is no information whether it is effective in obese individuals or not. Also, it should be clarified if obesity influences response to periodontal treatment. This study hypothesized that obesity impair response to periodontal treatment. Therefore, the effects of the protocol "one-stage full-mouth disinfection" will be evaluated in obese individuals and normal weight controls. This evaluation will be based on the monitoring of several clinical, microbiological and biochemical parameters throughout 9 months. Participants will answer validated questionnaires to evaluate if treatment of gum disease would be able to improve individual's quality of life. Study population will be composed of 90 to 100 obese individuals (males or females; > 18 years of age; smokers or non smokers; > 12 natural teeth). Participants will be classified into 5 groups according to their body mass index in normal weight (n = 15 to 20); overweight (n = 15 to 20); obesity I (n = 15 to 20); obesity II (n = 15 to 20); obesity III (n = 15 to 20). Examinations will be performed before treatment and also 3, 6 and 9 months after treatment. This study will contribute to the knowledge on how obese individuals respond to this specific treatment protocol. Also, having normal weight individuals as controls the present study will contribute to a better understanding about obesity, in its different severities, influence on periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to advanced generalized chronic periodontitis
* Body mass index: > 18.5 kg/m2
* Minimum of 12 natural teeth
* Smokers, non-smokers or former-smokers

Exclusion Criteria:

* Systemic diseases (diabetes, renal diseases, rheumatic diseases, osteoporosis and cardiovascular diseases)
* Pregnant and lactating women
* HIV/ AIDS
* periodontal treatment in the last year (before baseline appointment)
* Medication: Immunosuppressive drugs, antibiotics in the past three months (before baseline appointment) )
* orthodontic appliance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Periodontal clinical efficacy | Changes in periodontal pocket depth measurements from baseline to 6 months
  Improvements in periodontal pocket depth (mm) overtime and comparisons among groups at 6 months after treatment
Periodontal clinical efficacy | Changes in clinical attachment measurements from baseline to 6 months
  Improvements in clinical attachment level (mm) overtime and comparisons among groups at 6 months after treatment

SECONDARY OUTCOMES:
Antimicrobial efficacy | Changes in total bacterial levels from baseline to 6 months
  Reductions in total bacterial levels and levels of target bacterial species overtime and comparisons among groups at 6 months after treatment
Antimicrobial efficacy | Changes in bacterial levels from baseline to 6 months
  Reductions in Treponema denticola, Porphyromonas gingivalis, Tannerella forsythia, Aggregatibacter actinomycetemcomitans levels overtime and comparisons among groups at 6 months after treatment
Oral safety and tolerability | Changes in salivary nitrite levels from baseline to 6 months
  Maintenance of salivary nitrite levels overtime and comparisons among groups at 6 months after treatment
Impact on quality of life | Changes in scores (Likert scale ranging from 16 to 80 points) of Oral health and quality of life - United Kingdom questionnaire from baseline to 6 months
  Improvements in Oral health and quality of life - United Kingdom questionnaire scores overtime and comparisons among groups at 6 months after treatment
Impact on quality of life | Changes in scores (Likert scale ranging from 0 to 56 points) of Oral impacts on daily performance questionnaire from baseline to 6 months
  Improvements in Oral impacts on daily performance questionnaire scores overtime and comparisons among groups at 6 months after treatment

OTHER OUTCOMES:
Systemic effects | Changes in in glycemic levels from baseline to 6 months.
  Glycemic blood levels.
Systemic effects | Changes in blood levels of high density lipoprotein-cholesterol, low density lipoprotein -cholesterol and very low density lipoprotein - fractions from baseline to 6 months.
  Blood levels of high density lipoprotein-cholesterol, low density lipoprotein -cholesterol, very low density lipoprotein - fractions levels parameters.
Systemic effects | Changes in blood counts of white cells, red cells and platelets from baseline to 6 months.
  Blood counts of white cells, red cells and platelets.

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Cortelli, PhD, Principal Investigator — Associate professor
Locations (1):
- University of Taubate, Taubaté, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared